CLINICAL TRIAL: NCT01110226
Title: Phase I Trial Of Cisplatin And KML-001 In Advanced Non-Small Cell Lung Cancer and Other Platinum Responsive Malignancies
Brief Title: Trial Of Cisplatin And KML-001 in Platinum Responsive Malignancies
Acronym: 0805GCC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity was not felt to be acceptable for further development.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040420; GCC 0805 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2009-12-14; First posted 2010-04-26 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Non-Small Cell Lung Cancer, Small Cell Lung Cancer; Platinum Responsive Malignancies
Keywords: non small cell lung cancer; small cell lung cancer; Platinum Responsive; solid tumor malignancies
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — sodium arsenite; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Period 1: KML001 15mg plus Cisplatin 75mg/m2 (Experimental): KML001 15 mg orally daily days 1-14 with cisplatin IV on day1
  Interventions: Drug: KML-001; Drug: Cisplatin
- Period 2: KML001 17.5mg plus Cisplatin 75mg/m2 (Experimental): KML001 17.5 mg orally daily days 1-14 with cisplatin IV on day1
  Interventions: Drug: KML-001; Drug: Cisplatin
- Period 3: KML001 20mg plus Cisplatin 75mg/m2 (Experimental): KML001 20 mg orally daily days 1-14 with cisplatin IV on day1
  Interventions: Drug: KML-001; Drug: Cisplatin

INTERVENTIONS:
Drug: KML-001 — KML001 will begin given to patients first. It should be taken by mouth immediately prior to cisplatin infusion. Patients will be treated in cohorts of three beginning at 15mg. The Dose will be increased until Maximum Tolerated Dose is established.
  KML001 will be administered daily for 14 days of a 21 day cycle. Patients will have one week off.
  Other Names: sodium metaarsenite
Drug: Cisplatin — Cisplatin will be given to all patients at a dose of 75 mg/m2 on day 1 of every 21 day cycle over 30 to 90 minutes through an intravenous infusion immediately after the first dose of KML-001

SUMMARY:
This is a Phase I Clinical Trial. Phase I studies are designed to determine the amount of investigational drugs that can be safely tolerated and to define the side effects that limit the dose. The drug administered in this study is KML-001. It is a highly soluble, orally available arsenic agent. It is currently being tested to determine its effects on telomerase activity.

In other words, the purpose of this research study is to find the highest dose of KML001, that can be given without causing severe side effects when it is combined with a standard, commercially available anti-cancer drug called cisplatin.

DETAILED DESCRIPTION:
Telomerase is the enzyme synthesizing the specific DNA sequences found at the telomeres in the body's chromosomes. It is thus responsible for maintaining the length of telomeres. Telomerase has been detected in human cancer cells and is found to be 10-20 times more active than in normal body cells. This provides a selective growth advantage to many types of tumors. If telomerase activity was to be turned off, then telomeres in cancer cells would shorten, just like they do in normal body cells. This would prevent the cancer cells from dividing uncontrollably in their early stages of development. In the event that a tumor has already thoroughly developed, it may be removed and anti-telomerase therapy could be administered to prevent relapse.

This study is being offered to patients with advanced cancer which has either no standard therapy or which has progressed after treatment with one or more standard treatments.

The primary objective of this study :

To determine the maximum tolerated dose of KML001 in combination with cisplatin in patients with advanced malignancy. This objective has been met. The study will be reopened with expansion cohorts in advanced small cell lung cancer and non-small cell lung cancer to better assess the activity of the combination, pending (Institutional Review Board (IRB) approval.

Secondary Objectives of the study:

To determine the pharmacokinetics of KML001 and cisplatin in this combination. To assess the response rate, disease-free survival and survival associated with this regimen.

To correlate indications of patient benefit (response or stable disease) with pretreatment specimens

The highest safest doses are determined by increasing the doses of cisplatin and KML001 in successive groups of patients until at least some of them have serious side effects. All patients on this study will receive the same dose of cisplatin, which is known to have antitumor effects. The doses of KML001 will be increased in successive groups of patients. It is possible that those entering the study early may receive suboptimal doses of KML001. At the end of the study we hope to determine the appropriate dose of the KML001 in combination with cisplatin, learn about its side effects and understand how the body metabolizes the drug.

Laboratory data from the University of Maryland Greenebaum Cancer Center (UMGCC) has demonstrated that the combination of KML001 and cisplatin is synergistic in lung cancer cell lines. Cisplatin is the best established agent for the treatment of lung cancer and most treatment regimens have been established with cisplatin (or its congener, carboplatin). This synergism is particularly interesting given that there is an anti-telomere effect for cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer or other "platinum responsive malignancies" , including but not limited to: esophageal cancer, ovarian cancer, germ cell malignancies , transitional cell cancer etc. that are not curable with chemotherapy, surgery or radiotherapy. A tissue block or fresh tissue biopsy is required. Patients with CNS (Central Nervous System) metastases which are symptomatic must have received therapy (surgery, X Ray Therapy (XRT), gamma knife) and be neurologically stable and off steroids. Patients with asymptomatic lesions without significant edema and no evidence of shift are allowed to participate without prior CNS therapy. Such patients are anticipated to receive specific CNS therapy after 2-4 courses of therapy.
* Patients may have received prior systemic chemotherapy or radiation therapy. At least 2 weeks should have elapsed since the last treatment and patients should have recovered from previous significant toxicity (i.e. to grade 1 or less). Alopecia, skin discoloration etc. are not considered significant toxicities. There is no limit on the number of prior therapies. Patients may have received prior cisplatin or other platinum regimens.
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.
* Patient 18 years of age or older.
* Absolute Granulocyte Count greater than or equal to 1.5 x 10^9
* Platelet count greater than or equal to 100 x 10^9
* Serum creatinine within normal limits, or an estimated or measured creatinine clearance greater than or equal to 65 ml/min.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent.
* Serum calcium, magnesium and potassium must be within normal limits.

Exclusion Criteria:

* Patients must not have serious infection or other serious underlying medical condition which would impair the ability of the patient to receive protocol treatment. These need not be specified in the history and physical and can be documented through signature on the eligibility checklist. Severe, active co-morbidity, defined as follows:

  1. Current uncontrolled cardiac disease;
  2. Corrected (Bazett) QTc interval of > .50 ms (male) or > .52 ms (female);
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 4 weeks of registration;
  5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
  6. Patients with acquired Immune Deficiency Syndrome (AIDS) based upon current Center for Disease Control (CDC) definition or patients known to be HIV positive.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* Pre-existing ≥ grade 2 peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2015-10-22 (Actual); Study Completion 2015-10-27 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of KML001 in combination with cisplatin | DLT to be determined up to 30 days after administration
  Once 3 subjects in a cohort reach a dose limiting toxicity. In this protocol, it took 23 months to determine the dose limiting toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Edelman, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phatak P, Dai F, Butler M, Nandakumar MP, Gutierrez PL, Edelman MJ, Hendriks H, Burger AM. KML001 cytotoxic activity is associated with its binding to telomeric sequences and telomere erosion in prostate cancer cells. Clin Cancer Res. 2008 Jul 15;14(14):4593-602. doi: 10.1158/1078-0432.CCR-07-4572. PMID 18628474